CLINICAL TRIAL: NCT02582112
Title: Do Warming iv Fluids During the Management of Spinal- Induced Hypotension Decrease the Incidence of Hypotension and Reduce the Requirement of Fluid, Blood and Ephedrine?
Brief Title: Warming IV Fluids and Incidence of Hypotension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hakki Unlugenc (Other)
Responsible Party: Sponsor-Investigator, Hakki Unlugenc, Professor Dr, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HZLTNS98
Record Dates: First submitted 2015-10-14; First posted 2015-10-21 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Assault by Hot Fluids

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warming group (Active Comparator): Active Comparator: Warming group
  Interventions: Other: Active Comparator: Warming group
- Control group (Placebo Comparator): Control group
  Interventions: Other: Active Comparator: Warming group

INTERVENTIONS:
Other: Active Comparator: Warming group — Placebo Comparator: Control group

SUMMARY:
This prospective, double-blinded, randomized, controlled study was undertaken to evaluate whether warming IV fluids (37 oC) resulted in lower incidence of hypotension, less ephedrine and transfusion requirement and lower fluid consumption than use of room-temperature fluids (22 oC) in cesarean delivery patients undergoing spinal anesthesia.

DETAILED DESCRIPTION:
Inadvertent perioperative hypothermia during cesarean delivery is not rare and frequently neglected, despite the recommendations by clinical guidelines. Exposure to cold air and infusing non-warmed intravenous (iv) fluids are the other main sources of inadvertent hypothermia. Spinal anesthesia used during the cesarean delivery has also been demonstrated to impair normal autonomic thermoregulatory control and extend inadvertent perioperative hypothermia. Various measures such as pre-warming of patients or fluids before anesthesia, peroperative warming of iv fluids and active/passive cutaneous warming techniques have all been used to prevent or to reduce inadvertent perioperative hypothermia. This prospective, double-blinded, randomized, controlled study was undertaken to evaluate whether warming IV fluids (37 oC) resulted in lower incidence of hypotension, less ephedrine and transfusion requirement and lower fluid consumption than use of room-temperature fluids (22 oC) in cesarean delivery patients undergoing spinal anesthesia.

The hypothesis was that in elective caesarean delivery patients undergoing spinal anesthesia, warming intravenous fluids, would reduce the incidence of hypotension, ephedrine and transfusion requirement and volume consumption. Thus, the primary outcome measure of the present study was the incidence of intraoperative maternal hypotension and ephedrine requirement during spinal anaesthesia for caesarean section. Secondary outcome measures were total volume consumption, blood loss, pain scores, shivering and maternal and foetal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were previous cesarean delivery and breech presentation.

Exclusion Criteria:

* Exclusion criteria included parturients younger than 18 and older than 43 years, significant coexisting disease such as preeclampsia or eclampsia, thyroid disorders, neurological disorders, increased risk of intra-operative hemorrhage (such as placenta accreta), and any contraindication to regional anaesthesia such as bleeding disorders or local infection.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the present study was the incidence of intraoperative maternal hypotension and ephedrine requirement during spinal anaesthesia for caesarean section | 6 months
  Systolic and diastolic blood pressures (mmHg) and Ephedrine and transfusion requirement (n /mg)

SECONDARY OUTCOMES:
Secondary outcome measures were total volume consumption. | 6 months
  Total volume consumption (mL),
Secondary outcome measures were pain scores | 6 months
  Pain scores (VRS),
Secondary outcome measures were shivering and maternal and foetal side effects. | 6 months
  side effects such as shivering, nausea, vomiting, bradycardia, hypoxia (y/n)

CONTACTS AND LOCATIONS:
Overall Officials: Hakkı Ünlügenç, Prof Dr, Study Director — Cukurova University
Locations (1):
- Hakki Unlugenc, Adana, Turkey (Türkiye)